CLINICAL TRIAL: NCT05221294
Title: Modified Del Nido Versus Custodiol Cardioplegia For Myocardial Protection In Adult Patients Undergoing Cardiac Surgery; A Prospective Randomized Double-Blinded Clinical Trial.
Brief Title: Modified Del Nido Versus Custodiol Cardioplegia For Myocardial Protection In Cardiac Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mahdy Ahmed Abd Elhady, Fayoum University Hospital, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R193
Record Dates: First submitted 2021-12-20; First posted 2022-02-02 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2022-10

CONDITIONS: Cardioplegia Solution Adverse Reaction
Keywords: Myocardial Protection; Custodiol Cardioplegia; Del Nido

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MDN group (Experimental): will receive modified Del Nido cardioplegia solution
  Interventions: Drug: Modified Del Nido Versus Custodiol Cardioplegia
- C group (Experimental): will receive Custodiol cardioplegia
  Interventions: Drug: Modified Del Nido Versus Custodiol Cardioplegia

INTERVENTIONS:
Drug: Modified Del Nido Versus Custodiol Cardioplegia — Modified Del Nido Versus Custodiol Cardioplegia For Myocardial Protection In Cardiac Surgery

SUMMARY:
Cardioplegia solutions have been considered as a corner stone for myocardial protection during cardiac surgery with cardiopulmonary bypass and cardiac arrest, it limits the metabolic activity and increases the capacity of the myocardium to withstand prolonged ischemic time, and thus it has a direct impact on surgical outcomes. (1, 2) Long acting cardioplegic solutions with a single dose strategy are beneficial as they allow surgery without interruptions, reducing cross clamp time and provide more cardiac protection. (3) Custodiol (histidine- tryptophan- ketoglutarate) solution has been described in the 1970s by Bretschneider (4), and used as an alternative to hyperkalemic crystalloid solutions especially during complex cardiac surgeries, also used for organ preservation during transplant surgery. (5, 6) In the 1990s Pedro del Nido and his team introduced a new cardioplegic solution (del Nido cardioplegia) for pediatric cardiac surgeries. (7) But recently, many studies postulated its use for adults. (8) The base solution for the traditional del Nido cardioplegia is Plasma-Lyte A which is a calcium free solution and electrolyte composition similar to the extracellular fluid. (7) However Plasma-Lyte A is unavailable in many countries, this precludes its use. Some authors have advocated lactated Ringer's as a base solution instead of Plasma-Lyte A for preparing del Nido cardioplegia, now known as modified del Nido cardioplegia. (9) Custodiol and modified del Nido cardioplegia can be used in a single dose fashion with proper myocardial protection and minimal surgical interruptions. However, the literature also does not confirm the superiority of one over another. (1) Also, limited number of clinical trials compared both cardioplegic solutions directly. So, in this study we aimed to assess the efficacy of both Custodiol and modified del Nido cardioplegia in myocardial protection and clinical outcomes among adult patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Patients will be divided into two groups with 1:1 allocation, randomized by computer generated random numbers that will be placed in separate opaque envelopes opened by study investigators at OR. MDN group (will receive modified Del Nido cardioplegia solution) and C group (will receive Custodiol cardioplegia). Participants and data collectors will be blinded with the group allocation till the end of the study.

Inclusion criteria: patients ≥ 18 years old, scheduled for elective valve replacement surgery or coronary artery bypass grafting surgery.

All patients will be preoperatively examined and investigated by complete blood count, coagulation profile, liver and kidney functions and electrolytes. Electrocardiography, chest x ray and echocardiography will be routinely done. Coronary angiography and carotid arterial duplex will be requested on demand.

Patient will be premedicated by intramuscular injection of 10mg morphine at morning of the operation. Before induction of anesthesia, a five-lead electrocardiography system will be applied to monitor heart rate, rhythm, and ST segments (leads II and V5). A pulse oximeter probe will be attached, and a peripheral venous cannula will be placed. For measurement of arterial pressure and blood sampling, a 20 G cannula will be inserted into either right or left radial artery under local anesthesia. After pre-oxygenation, general anesthesia will be induced by midazolam 2-5 mg, fentanyl (10μg/kg), propofol (3-4mg/Kg), followed by atracurium (0.5 mg/kg).

Trachea will be intubated; patients will be mechanically ventilated with oxygen in air so as to achieve normocarbia. This will be confirmed by radial arterial blood gas analysis and capnogram. An esophageal temperature probe and a urinary catheter will also be placed. For drug infusion, a triple-lumen central venous catheter will be inserted via the right internal jugular vein. Anesthesia will be maintained by inhaled Isoflurane 0.4 to 1% and atracurium infusion at a rate of 0.5 mg/kg/h for continued muscle relaxation. During extracorporeal circulation, patients will receive propofol infusion at a rate of 50-100 µ/kg/min. in addition to atracurium infusion.

Before initiation of cardiopulmonary bypass (CPB), the patients will receive intravenous heparin (300-500 units/kg body weight) to achieve an activated clotting time >480s. CPB will be instituted via an ascending aortic cannula and a two-stage right atrial cannula. Before, during (pump blood flow: 2.4l/min/m2), and after CPB, mean arterial pressure will be adjusted to exceed 60mmHg.

Surgery will be done via median sternotomy; CBP will be established via arterial cannula in the ascending aorta and venous drainage obtained via two-stage cannula in the right atrium or bicaval cannulation.

Myocardial protection:

Cardioplegic solution will be administered via antegrade technique through the aortic root or the coronary ostia accordingly. Patients will receive either Custodiol cardioplegia or modified Del Nido cardioplegia according to their allocation.

Ready Custodiol cardioplegia solution will be administered in a single dose of 25ml.kg-1 over 6-8 minutes with 4-8 oC temperature and 150-200 mmHg infusion pressure. Custodiol is a ready sterile cardioplegia composed of; sodium chloride 15 mmol/L, potassium chloride 9 mmol/L, magnesium chloride 4 mmol/L, calcium chloride 0.015 mmol/L, histidine 180 mmol/L, tryptophan 2 mmol/L, ketoglutarate 1 mmol/L and mannitol 30 mmol/L with pH 7.4-7.45 at 4°C and osmolality 310 mosmol/Kg.

Modified Del Nido cardioplegia will be prepared at OR, and lactated Ringer's solution will be used as a crystalloid base, with crystalloid: blood ratio of 4:1 and will be given with a dose of 20 ml/kg (with a maximum dose of 1000 ml) at 4 oC temperature and 200-300 mmHg administration pressure and if necessary additional dose will be given after 90 minutes of the initial dose. The composition of modified Del Nido cardioplegia will be as follows: lactated Ringer's solution 1000ml, 13 ml sodium bicarbonate (1 mEq/ ml), 16.3 ml of mannitol 20%, 4 ml magnesium 50%, 6.5 ml of lidocaine 2% and 13ml of potassium chloride (2 mEq/L).

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years old, scheduled for elective valve replacement surgery or coronary artery bypass grafting surgery.

Exclusion Criteria:

* Emergency surgery.
* Chronic kidney disease.
* Hepatic impairment.
* Re-do surgery.
* Severe psychiatric illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
troponin I | 24 hours after surgery
  troponin I at 24 hours after surgery to assess myocardial protection between the two used cardioplegia solutions.

SECONDARY OUTCOMES:
The total volume of cardioplegia solution | In the first 24 hours of surgery
  The total volume of cardioplegia solution
Total cross-clamp time and total CPB time | In the first 24 hours of surgery
  Total cross-clamp time and total CPB time
Incidence of ventricular fibrillation after cross-camp removal | In the first 24 hours of surgery
  side effects
Postoperative left ventricular ejection fraction | 24 hours after surgery in days
  Postoperative left ventricular ejection fraction
Requirement of inotropes and time of discontinuation | postoperative 24 hours
  intraoperative
Troponin I at 12 hours after surgery | postoperative 24 hours
  Troponin I at 12 hours after surgery
CK-MB at 12 and 24 hours after surgery | 24 hours after surgery
  assessment
Serum lactate level at 24 hours after surgery. | 24 hours after surgery
  assessment
Incidence of postoperative AF and MI. | 24 hours after surgery
  assessment
Time for weaning from mechanical ventilation | 24 hours after surgery in hours
  Time for weaning from mechanical ventilation
ICU length of stay | 24 hours after surgery in days
  assessment
hospital length of stay | 24 hours after surgery in days
  assessment

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hamed, M.D, Study Director — Fayoum University Hospital
Locations (1):
- Fayoum University hospital, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sanetra K, Pawlak I, Cisowski M. Del Nido cardioplegia - what is the current evidence? Kardiochir Torakochirurgia Pol. 2018 Jun;15(2):114-118. doi: 10.5114/kitp.2018.76477. Epub 2018 Jun 25. PMID 30069192
- [Result] Vivacqua A, Robinson J, Abbas AE, Altshuler JM, Shannon FL, Podolsky RH, Sakwa MP. Single-dose cardioplegia protects myocardium as well as traditional repetitive dosing: A noninferiority randomized study. J Thorac Cardiovasc Surg. 2020 May;159(5):1857-1863.e1. doi: 10.1016/j.jtcvs.2019.03.125. Epub 2019 May 11. PMID 31204129
- [Derived] Abdelhady MA, Goda AS, Sayed Gomaa MS, Hamed MA, Hassan AASM. Modified Del Nido Versus Custodiol(R) Cardioplegia for Myocardial Protection in Adult Patients Undergoing Cardiac Surgery; A Prospective Randomized Double-Blinded Clinical Trial. Ann Card Anaesth. 2025 Oct 1;28(4):451-458. doi: 10.4103/aca.aca_35_25. Epub 2025 Oct 13. PMID 41081689